CLINICAL TRIAL: NCT00370214
Title: REVEAL Registry™: Registry to Evaluate Early And Long-term PAH Disease Management
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: CR001
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary arterial hypertension; Lung diseases; Heart diseases; Pulmonary circulation; Vascular resistance; PAH; Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Lung Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The REVEAL Registry™ is a multicenter, observational, U.S.-based study of the clinical course and disease management of pulmonary arterial hypertension (PAH) patients. All consecutive consenting patients diagnosed with WHO Group I PAH according to specific hemodynamic criteria at participating institutions will be enrolled. Participating patients will be followed for a minimum of five years from the time of enrollment.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a chronic, progressive, and often fatal disease characterized by severe constriction of the blood vessels in the lungs. Over the past decade, significant strides have been made in the medical management and understanding of PAH. However, much remains to be learned about the clinical course of both idiopathic PAH and associated PAH, including clinical presentation, pace of progression, key parameters to monitor, impact of treatment, and prognosticators of outcome. As the unique body of knowledge generated by the REVEAL Registry grows, it is hoped that new understandings, insights, and treatments will emerge that will improve the lives of patients with PAH.

The REVEAL Registry will provide investigators with descriptive data regarding the clinical course and treatment outcomes in patients with WHO Group I PAH. Data derived from the study may offer important tools for assessing current management practices of treating investigators, as well as changes over time. Additionally, the relationship of patient- and disease-specific parameters to patient outcomes may be able to be assessed through analysis of data from this study.

The specific objectives of the REVEAL Registry™ are to:

* Characterize the demographics and clinical course of PAH patients
* Evaluate and compare patient outcomes
* Identify clinical predictors of short-term and long-term clinical outcomes
* Assess the relationship between PAH medications and patient outcomes
* Report temporal trends in treatments and outcomes for newly diagnosed patients
* Collect timely and relevant data for the evolving research needs of the PAH community

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or previously diagnosed patients with WHO Group I PAH.
* Documentation of the following hemodynamic parameters by right heart catheterization, performed at any time prior to study enrollment:
* Mean pulmonary arterial pressure (mPAP) >25 mm Hg at rest or mPAP > 30 mm Hg with exercise contemporaneous with a pulmonary wedge pressure ≤ 18 mm Hg
* Pulmonary wedge pressure ≤ 18 mm Hg
* Pulmonary vascular resistance (PVR) ≥ 240 dynes.sec.cm-5 (i.e., ≥ 3.0 Wood units)

Exclusion Criteria:

* Patients who meet the criteria for inclusion into WHO Groups II, III, IV or V
* Have not had documentation of hemodynamic criteria for PAH by right heart catheterization at some time preceding study entry and following development of symptoms associated with PAH.
* Do not meet the required hemodynamic criteria for entry into the study

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with WHO Group I Pulmonary Arterial Hypertension from US based PAH centers.
Sampling Method: Probability Sample
Enrollment: 3515 (Actual)
Dates: Start 2006-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Survival | 5 years

SECONDARY OUTCOMES:
clinical predictors, precise outcome definitions | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. McGoon, M.D., Study Chair — Mayo Clinic - Rochester, Minnesota; David B. Badesch, M.D., Study Director — University of Colorado, Denver; Robyn J. Barst, M.D., Study Director — Columbia University; Raymond Benza, M.D., Study Director — University of Alabama at Birmingham; Gregory Elliott, M.D., Study Director — LDS Hospital; Harrison Farber, M.D., Study Director — Boston Medical Center; Adaani Frost, M.D., Study Director — Baylor College of Medicine; Abby Krichman, RRT, Study Director — Duke University Pulmonary Vascular Disease Center
Locations (54):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Medical Center, Tucson, Arizona
  - University of California, San Diego, La Jolla, California
  - UCLA / VA Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Univeristy of California, San Francisco - Division of Cardiology and Pediatric ICU, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - UCLA School of Medicine: Harbor-UCLA, Torrance, California
  - The Children's Hospital, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Suncoast Lung Center, Sarasota, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - Midwest Heart Foundation, Naperville, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Kentucky Pulmonary Associates, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Children's Hospital, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Legacy Pulmonary Hypertension Clinic, Portland, Oregon
  - Penn Presbyterian Medial Center, Philadelphia, Pennsylvania
  - Temple Lung Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University Texas Health Science Center, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Benza RL, Kanwar MK, Raina A, Scott JV, Zhao CL, Selej M, Elliott CG, Farber HW. Development and Validation of an Abridged Version of the REVEAL 2.0 Risk Score Calculator, REVEAL Lite 2, for Use in Patients With Pulmonary Arterial Hypertension. Chest. 2021 Jan;159(1):337-346. doi: 10.1016/j.chest.2020.08.2069. Epub 2020 Sep 1. PMID 32882243
- [Derived] Torbicki A, Bacchi M, Delcroix M, Farber HW, Ghofrani HA, Hennessy B, Jansa P, Mehta S, Perchenet L, Pulido T, Rosenberg D, Rubin LJ, Sastry BKS, Simonneau G, Sitbon O, Souza R, Wei LJ, Channick R, Benza R. Integrating Data From Randomized Controlled Trials and Observational Studies to Assess Survival in Rare Diseases. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005095. doi: 10.1161/CIRCOUTCOMES.118.005095. PMID 31109190
- [Derived] Benza RL, Gomberg-Maitland M, Elliott CG, Farber HW, Foreman AJ, Frost AE, McGoon MD, Pasta DJ, Selej M, Burger CD, Frantz RP. Predicting Survival in Patients With Pulmonary Arterial Hypertension: The REVEAL Risk Score Calculator 2.0 and Comparison With ESC/ERS-Based Risk Assessment Strategies. Chest. 2019 Aug;156(2):323-337. doi: 10.1016/j.chest.2019.02.004. Epub 2019 Feb 14. PMID 30772387
- [Derived] Preston IR, Roberts KE, Miller DP, Sen GP, Selej M, Benton WW, Hill NS, Farber HW. Effect of Warfarin Treatment on Survival of Patients With Pulmonary Arterial Hypertension (PAH) in the Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL). Circulation. 2015 Dec 22;132(25):2403-11. doi: 10.1161/CIRCULATIONAHA.115.018435. Epub 2015 Oct 28. PMID 26510696
- [Derived] Farber HW, Miller DP, Poms AD, Badesch DB, Frost AE, Muros-Le Rouzic E, Romero AJ, Benton WW, Elliott CG, McGoon MD, Benza RL. Five-Year outcomes of patients enrolled in the REVEAL Registry. Chest. 2015 Oct;148(4):1043-54. doi: 10.1378/chest.15-0300. PMID 26066077
- [Derived] Chung L, Farber HW, Benza R, Miller DP, Parsons L, Hassoun PM, McGoon M, Nicolls MR, Zamanian RT. Unique predictors of mortality in patients with pulmonary arterial hypertension associated with systemic sclerosis in the REVEAL registry. Chest. 2014 Dec;146(6):1494-1504. doi: 10.1378/chest.13-3014. PMID 24992469
- [Derived] Burger CD, Long PK, Shah MR, McGoon MD, Miller DP, Romero AJ, Benton WW, Safford RE. Characterization of first-time hospitalizations in patients with newly diagnosed pulmonary arterial hypertension in the REVEAL registry. Chest. 2014 Nov;146(5):1263-1273. doi: 10.1378/chest.14-0193. PMID 24901386
- [Derived] Frost AE, Badesch DB, Miller DP, Benza RL, Meltzer LA, McGoon MD. Evaluation of the predictive value of a clinical worsening definition using 2-year outcomes in patients with pulmonary arterial hypertension: a REVEAL Registry analysis. Chest. 2013 Nov;144(5):1521-1529. doi: 10.1378/chest.12-3023. PMID 23907471
- [Derived] Bersohn MM, Turner MP, Traiger GL, Frost AE, Shapiro S. Systemic BP and heart rate as prognostic indicators in pulmonary arterial hypertension. Chest. 2013 Sep;144(3):959-965. doi: 10.1378/chest.12-2572. PMID 23598723
- [Derived] Barst RJ, Chung L, Zamanian RT, Turner M, McGoon MD. Functional class improvement and 3-year survival outcomes in patients with pulmonary arterial hypertension in the REVEAL Registry. Chest. 2013 Jul;144(1):160-168. doi: 10.1378/chest.12-2417. PMID 23429998
- [Derived] Poms AD, Turner M, Farber HW, Meltzer LA, McGoon MD. Comorbid conditions and outcomes in patients with pulmonary arterial hypertension: a REVEAL registry analysis. Chest. 2013 Jul;144(1):169-176. doi: 10.1378/chest.11-3241. PMID 23348820
- [Derived] Kitterman N, Poms A, Miller DP, Lombardi S, Farber HW, Barst RJ. Bloodstream infections in patients with pulmonary arterial hypertension treated with intravenous prostanoids: insights from the REVEAL REGISTRY(R). Mayo Clin Proc. 2012 Sep;87(9):825-34. doi: 10.1016/j.mayocp.2012.05.014. Epub 2012 Aug 9. PMID 22883740
- [Derived] Frost AE, Farber HW, Barst RJ, Miller DP, Elliott CG, McGoon MD. Demographics and outcomes of patients diagnosed with pulmonary hypertension with pulmonary capillary wedge pressures 16 to 18 mm Hg: insights from the REVEAL Registry. Chest. 2013 Jan;143(1):185-195. doi: 10.1378/chest.11-1387. PMID 22661451
- [Derived] Benza RL, Miller DP, Barst RJ, Badesch DB, Frost AE, McGoon MD. An evaluation of long-term survival from time of diagnosis in pulmonary arterial hypertension from the REVEAL Registry. Chest. 2012 Aug;142(2):448-456. doi: 10.1378/chest.11-1460. PMID 22281797
- [Derived] Barst RJ, McGoon MD, Elliott CG, Foreman AJ, Miller DP, Ivy DD. Survival in childhood pulmonary arterial hypertension: insights from the registry to evaluate early and long-term pulmonary arterial hypertension disease management. Circulation. 2012 Jan 3;125(1):113-22. doi: 10.1161/CIRCULATIONAHA.111.026591. Epub 2011 Nov 15. PMID 22086881
- [Derived] Krowka MJ, Miller DP, Barst RJ, Taichman D, Dweik RA, Badesch DB, McGoon MD. Portopulmonary hypertension: a report from the US-based REVEAL Registry. Chest. 2012 Apr;141(4):906-915. doi: 10.1378/chest.11-0160. Epub 2011 Jul 21. PMID 21778257
- [Derived] Shapiro S, Traiger GL, Turner M, McGoon MD, Wason P, Barst RJ. Sex differences in the diagnosis, treatment, and outcome of patients with pulmonary arterial hypertension enrolled in the registry to evaluate early and long-term pulmonary arterial hypertension disease management. Chest. 2012 Feb;141(2):363-373. doi: 10.1378/chest.10-3114. Epub 2011 Jul 14. PMID 21757572
- [Derived] Benza RL, Gomberg-Maitland M, Miller DP, Frost A, Frantz RP, Foreman AJ, Badesch DB, McGoon MD. The REVEAL Registry risk score calculator in patients newly diagnosed with pulmonary arterial hypertension. Chest. 2012 Feb;141(2):354-362. doi: 10.1378/chest.11-0676. Epub 2011 Jun 16. PMID 21680644
- [Derived] Brown LM, Chen H, Halpern S, Taichman D, McGoon MD, Farber HW, Frost AE, Liou TG, Turner M, Feldkircher K, Miller DP, Elliott CG. Delay in recognition of pulmonary arterial hypertension: factors identified from the REVEAL Registry. Chest. 2011 Jul;140(1):19-26. doi: 10.1378/chest.10-1166. Epub 2011 Mar 10. PMID 21393391
- [Derived] Burger CD, Foreman AJ, Miller DP, Safford RE, McGoon MD, Badesch DB. Comparison of body habitus in patients with pulmonary arterial hypertension enrolled in the Registry to Evaluate Early and Long-term PAH Disease Management with normative values from the National Health and Nutrition Examination Survey. Mayo Clin Proc. 2011 Feb;86(2):105-12. doi: 10.4065/mcp.2010.0394. PMID 21282484
- [Derived] Benza RL, Miller DP, Gomberg-Maitland M, Frantz RP, Foreman AJ, Coffey CS, Frost A, Barst RJ, Badesch DB, Elliott CG, Liou TG, McGoon MD. Predicting survival in pulmonary arterial hypertension: insights from the Registry to Evaluate Early and Long-Term Pulmonary Arterial Hypertension Disease Management (REVEAL). Circulation. 2010 Jul 13;122(2):164-72. doi: 10.1161/CIRCULATIONAHA.109.898122. Epub 2010 Jun 28. PMID 20585012
- [Derived] Frost AE, Badesch DB, Barst RJ, Benza RL, Elliott CG, Farber HW, Krichman A, Liou TG, Raskob GE, Wason P, Feldkircher K, Turner M, McGoon MD. The changing picture of patients with pulmonary arterial hypertension in the United States: how REVEAL differs from historic and non-US Contemporary Registries. Chest. 2011 Jan;139(1):128-37. doi: 10.1378/chest.10-0075. Epub 2010 Jun 17. PMID 20558556
- [Derived] Chung L, Liu J, Parsons L, Hassoun PM, McGoon M, Badesch DB, Miller DP, Nicolls MR, Zamanian RT. Characterization of connective tissue disease-associated pulmonary arterial hypertension from REVEAL: identifying systemic sclerosis as a unique phenotype. Chest. 2010 Dec;138(6):1383-94. doi: 10.1378/chest.10-0260. Epub 2010 May 27. PMID 20507945
- See also: Official REVEAL Registry website — http://www.REVEALregistry.com
- See also: PAH clinical studies at Mayo Clinic — http://www.mayoclinic.org/pulmonary-hypertension/clintrials.html